CLINICAL TRIAL: NCT00111332
Title: Exercise Effects in HIV-Infected Women
Brief Title: Study of Home-Based Resistance and Strength Training in HIV-Infected Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49302-P2 (completed); R01DK049302 (NIH)
Record Dates: First submitted 2005-05-19; First posted 2005-05-20 (Estimated); Last update posted 2010-04-14 (Estimated); Status verified 2010-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Behavioral: Progressive resistance and aerobic training

SUMMARY:
Lipodystrophy is characterized by increased cardiovascular disease. Limited strategies are available to increase cardiovascular fitness in this population, particularly among women. Progressive aerobic and resistance training will increase aerobic capacity and improve strength in HIV positive women with lipodystrophy.

DETAILED DESCRIPTION:
Baseline Testing: Eligible patients will be tested at the General Clinical Research Center (GCRC) of Massachusetts General Hospital or at the GCRC at Massachusetts Institute of Technology (MIT). For women with regular menses, the admission will correspond to the early follicular phase. Patients will receive a menstrual history calendar to submit at the baseline and 16 week visits. A complete history and physical exam will be performed, including a detailed history of all drugs being used in the treatment of the HIV disease or any associated conditions. Weight will be measured and expressed as a percentage of ideal body weight (IBW) and body mass index. Blood will be sampled to determine hormonal function (testosterone, free testosterone, SHBG, estradiol, LH, and FSH), nutritional status (albumin, prealbumin), lipid parameters (HDL, LDL, cholesterol, triglycerides), immune function (CD4, viral load, CBC), and thrombolytic markers (t-PA, PAI-1). An HIV test will be performed at the baseline visit only, in order to document patient status. Glucose homeostasis will be measured with the use of fasting glucose and insulin levels and an oral glucose tolerance test (OGTT). Heart rate will be monitored to test cardiovascular function. A spot urine will be collected for bone markers and beta-human chorionic gonadotropin (bHCG). Lean body mass and fat mass will be determined by a dual energy x-ray absorptiometry [DEXA] (to be performed at the MIT CRC); total body water will be determined by bioimpedance analysis; muscle cross-sectional area will be determined by anthropometric measurements. A quantitative computed tomography (CT) scan of the thigh and abdomen will be done to measure visceral and subcutaneous fat. A Magnetic Resonance Spectroscopy of calf muscles for determination of lipid concentrations in skeletal muscle will be done. (Subjects with contraindications to magnetic resonance imaging [MRI] will be able to remain in the protocol, but the MR-Spectroscopy will not be performed). A complete dietary assessment and resting energy expenditure will be performed. Quality of life will be assessed using the MOS HIV questionnaire and an activity questionnaire as well as the Karnofsky performance assessment.

A submaximal exercise bicycle test will be done to assess aerobic capability, and a 6 minute walk test, sit to stand and get up and go tests will be done to assess overall functional status by the physical therapy (PT) department. Those who are not randomized to exercise at the baseline visit, will have one repetition maximum (1 RM) testing. The 1 RM is defined as the maximal amount of weight that can be lifted throughout full range of motion. The 1 RM will be tested by performing exercises including calf raises, arm curls, lateral raises, knee flexors, bench press and half squats. The 1 RM testing will be repeated on those who are not randomized to exercise at the 8 and 16 week visits.

After the baseline investigation is over, subjects will be randomized into one of two groups (exercise or no exercise) for 16 weeks. Strength training will be performed using standard free weights under the supervision of a trained physical therapist or member of the study staff. Each session begins with a 5 minute warm-up and a standard flexibility routine. The strength training routine will follow and will focus on the following muscle groups: knee extensors and hip extensors, ankle plantar flexors, elbow flexors, pectoralis and shoulder abduction. The aerobic training program will follow the general guidelines established by the American College of Sports Medicine. Training will be performed using a standard stationery bicycle. Aerobic/endurance exercise will be performed with large muscle groups. The duration of the aerobic component of the training session will be 20 minutes during the first two weeks and 30 minutes thereafter. The intensity of the exercise will be 60% of maximal heart rate during the first two weeks and 75% thereafter. As the weeks progress, the repetitions and intensity of the exercise will be gradually increased. Subjects return to the GCRC at 8 weeks for a medical history, a physical exam, weight, and pregnancy test. Subjects return again at 16 weeks for a visit identical to that at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with documented HIV infection, by Western blot or ELISA
* Ages 18-60
* Self-report AND physical evidence, as assessed by the investigators, of at least one of the following:

  * increased abdominal girth;
  * relative loss of fat in the face;
  * relative loss of fat in the extremities; *dorsocervical fat pad;
  * relative increased breast size;
  * a score greater than or equal to 1.5 on the Lipodystrophy Scale and a waist to hip ratio of greater than or equal to 0.85.

Exclusion Criteria:

* Pregnant or actively seeking pregnancy
* Breastfeeding
* New opportunistic infection diagnosed within 4 weeks of the study
* Pharmacologic glucocorticoid therapy (> 7.5 mg Prednisone or its equivalent/day)
* Androgen, growth hormone or Megace within 3 months of study initiation
* New anti-retroviral therapy within 1 month of the study
* SGOT > 5x normal and/or clinically significant liver disease
* Creatinine > 2.0 mg/dL and/or clinically significant renal disease
* Hemoglobin (Hgb) < 8.0g/dL
* Active substance abuse

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40
Dates: Start 2002-11; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
aerobic fitness

SECONDARY OUTCOMES:
strength
body composition
lipids
glucose
cardiovascular disease (CVD) risk markers

CONTACTS AND LOCATIONS:
Locations (1):
- Mass General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Dolan SE, Frontera W, Librizzi J, Ljungquist K, Juan S, Dorman R, Cole ME, Kanter JR, Grinspoon S. Effects of a supervised home-based aerobic and progressive resistance training regimen in women infected with human immunodeficiency virus: a randomized trial. Arch Intern Med. 2006 Jun 12;166(11):1225-31. doi: 10.1001/archinte.166.11.1225. PMID 16772251